CLINICAL TRIAL: NCT06062173
Title: Preoperative Prediction of Adherent Perirenal Fat Based on CT Radiomics Combined With Deep Learning: a Prospective, Multicenter Study.
Brief Title: Preoperative Prediction of Adherent Perirenal Fat.
Acronym: APF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: wangyanbo
Record Dates: First submitted 2023-08-29; First posted 2023-10-02 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-06

CONDITIONS: Radiomics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adherent perirenal fat group: The surgeon considers perirenal fat to be adherent.
- Non-adherent perirenal fat group: Perirenal fat is considered nonadherent by surgeons.

SUMMARY:
In addition to kidney tumor specific factors, adherent perirenal fat is one of the most important causes of technical complications in kidney surgery, and currently, there is a lack of widely used non-invasive predictive models in clinical practice. In this study, a deep learning algorithm based on CT imaging and nomogram was proposed to identify and predict the presence of adherent perirenal fat. This study includes the construction of a prediction model based on CT imaging and the verification of the prediction model.

DETAILED DESCRIPTION:
Importance:

For patients with kidney tumors requiring surgical treatment, adhesive perirenal fat is a frustrating variable that surgeons encounter during surgery, but the current image-dependent kidney morphometric scoring system used to predict the potential difficulty of surgery ignores this factor. Accurate preoperative prediction of perirenal fat status remains an urgent need.

Purpose:

To determine whether radiomics features of perirenal fat derived from computed tomography images can provide valuable information for judging perirenal fat status, develop a prediction model based on CT radiomics combined with deep learning, and validate the performance of the model in an independent cohort.

Design, setup and participants:

The study included one retrospective dataset and one prospective dataset from four medical centers between January 2020 and September 2023. Kidney plain CT scan was performed in xx adult patients with partial nephrectomy or radical nephrectomy. The training set, validation set, and internal test set were provided by the First Hospital of Jilin University, and the external test set was provided by the First Hospital of Siping City, Liaoyuan Central Hospital and Dongfeng County Hospital. This diagnostic study used single-institution data from January 2020 to May 2023 to extract imaging omics features from the perirenal fat region (independent sample T-test, minimum absolute contraction, and selection operator logistic regression was used to screen for the best imaging omics features). Univariate and multivariate analyses of clinical variables in patients prior to renal surgery were performed to determine independent predictors of adherent perirenal fat in the clinical setting. Different classifiers were used to build prediction models using only the image-omics features and fusion prediction models using independent clinical predictors combined with the image-omics features. Its performance is verified in two test sets.

Main achievements and measures:

The discriminant performance of the image omics model was evaluated by the area under the receiver operating characteristic curve and confirmed by decision curve analysis.

ELIGIBILITY:
Inclusion Criteria:

* （1）Renal tumors, patients requiring surgical treatment. (2) Patients with complete preoperative CT image data.

Exclusion Criteria:

-(1) Preoperative complications such as acute urinary tract infection, hydronephrosis, pulmonary infection, autoimmune disease, and blood system disease.

(2) Severe respiratory movement artifacts in CT images. (3) Pregnant or breastfeeding women. (4) Patients who have received immunotherapy or chemoradiotherapy.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Preoperative renal CT plain scan imaging data and related clinical data of patients who underwent partial nephrectomy or radical nephrectomy in the First Hospital of Jilin University from January 2022 to December 2022 were retrospectively collected. Imaging data and clinical data from other research centers from June 2023 to September 2023 were prospectively collected. Select the required data according to the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-01-05 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Radiomics features | From January 2020 to December 2023.
  Radiomics features related to the prediction of adherent perirenal fat.

CONTACTS AND LOCATIONS:
Overall Officials: yanbo wang, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- Yanbowang, Ch’ang-ch’un, Jilin, China